CLINICAL TRIAL: NCT04861181
Title: Study of the Relationship(s) Between Clinical, Biological and Pharmacokinetic Metrics and Toxicities When Niraparib is Used as Maintenance Treatment (300mg or 200 mg/Day) for Ovarian Cancer Patients.
Brief Title: NIRAPK : Study of the Relationship(s) Between Clinical, Biological and Pharmacokinetic Metrics and Toxicities When Niraparib is Used as Maintenance Treatment for Ovarian Cancer Patients.
Acronym: NIRAPK
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: End of inclusion period.
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 69HCL20_0989
Record Dates: First submitted 2021-04-20; First posted 2021-04-27 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Adult Patients With Platinum-sensitive, Relapsed, High Grade Serous Epithelial Ovarian Cancer
Keywords: Niraparid; Pharmacokinetic; Hematologic toxicity; Nephrotoxicity; Thrombocytopenia; Maintenance treatment; Ovarian cancer; Predictive factors
MeSH Terms: conditions — Recurrence; Thrombocytopenia; Ovarian Neoplasms | interventions — Pharmacokinetics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pharmacokinetics, Dosage of Niraparib (Experimental): Patients received 3 cycles of Niraparib (200 mg or 300 mg/day). Each cycle lasts 28 days. Serum niraparib assays will be performed for all patients over 3 courses immediately prior to treatment (Cycle 1 Day 1, Cycle 1 Day 15, Cycle 2 Day 1 and Cycle 3 Day 1). Close-up kinetic measurements will also be taken at 1 Hour, 2 Hours, 4 Hours, 6 Hours and 24 Hours at Cycle 1 Day 15.
  Interventions: Biological: Pharmacokinetics, Dosage of Niraparib

INTERVENTIONS:
Biological: Pharmacokinetics, Dosage of Niraparib — The biological samples collected during the NIRAPK study will be blood only. The complete biological work-up will be processed in the same way as the usual routine care procedure. Serum niraparib will be measured over 3 courses just prior to treatment (Cycle 1 Day 1, Cycle 1 Day 15, Cycle 2 Day 1 and Cycle 3 Day 1). Close-up kinetic measurements will also be taken at 1 Hour, 2 Hours, 4 Hours, 6 Hours and 24 Hours at Cycle 1 Day 15.

SUMMARY:
Ovarian cancer is the seventh most common cancer in women worldwide and is the leading cause of gynecologic cancer deaths in high-income countries.

Standard treatment for newly diagnosed advanced ovarian cancer consist of cytoreductive surgery and platinum-based chemotherapy with or without concurrent and maintenance bevacizumab, a vascular endothelial growth factor (VEGF) inhibitor.

A majority of women with epithelial ovarian cancer respond well to first-line platinum-based chemotherapy. There is however a high rate of relapse/recurrence (disease progression ranging from 10 to 26 months).

Poly ADP ribose polymerase inhibitors (PARPi), a new class of therapeutic molecules have recently revolutionized this paradigm, demonstrating progression-free survival (PFS) advantages in several trials.

The PARPi molecule Niraparib has obtained its market authorization after the NOVA trial as second maintenance treatment line, irrespectively of patients' BRCA-mutated gene or HR status.

Since, results of the Phase III trial PRIMA, have demonstrated that Niraparib can also provided a significant PFS increase as first line maintenance treatment, for adult patients with platinum-sensitive, relapsed, high grade serous epithelial ovarian cancer who are in response (complete response or partial response) to platinum-based chemotherapy, irrespectively of their BRCA-mutated gene or HR status.

However, despite its high therapeutic potential, Niraparib at standard dose (200 or 300mg/day) is known to lead to hematologic toxicity and/or nephrotoxicity. This was demonstrated during the NOVA trial (the dose of Niraparib having to be reduced in 80% of the patients to reduce toxicity).

A retrospective study of the NOVA trial indicates that 2 predictive factors leading to hematologic toxicity were a weight <77kg and an initial platelet count <175 G/L. However, it seems more complex as 50% of patients with an initial weight between 58 and 77kg have not reported thrombocytopenia. Same for platelet count. Creatinine clearance below 60ml/min and an hypoalbuminemia <35 g/l have also been identified in another study as predictive factors to thrombocytopenia.

The inter-individual heterogeneity in terms of toxicity regarding Niraparib is high and still not well understood.

The aim of our study is therefore to better identify which clinical, biological and pharmacokinetic metrics can be considered as toxicity induction causes when Niraparib is used as maintenance treatment (200 or 300mg/day) for ovarian cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient Study Information and written informed consent
* Social Security Affiliation
* Patient > 18 years old.
* Ovarian, tubular or peritoneal high-grade epithelial carcinoma, histologically proven. Recommendation of a maintenance treatment with Niraparib at standard dose (200-300mg/day)
* Glomerular filtration rate with standardized serum creatinine values using CKD-EPI formula ≥ 30ml/min/1.73m2 (https://www.kidney.org/professionals/kdoqi/gfr_calculator)
* Normal liver function with bilirubin < 1.5N
* 6-8 weeks break between last chemotherapy and Niraparib treatment initiation.
* Patient with an effective birth control

Exclusion Criteria:

* Minor patient
* Patient not able to understand the aim of the study or under curatorship
* Low grade carcinoma
* Pregnant or breastfeeding patient
* Hypersensivity to an active substance present in niraparib

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The target population for this study is adult patients over 18 years of age with primary high-grade serous epithelial ovarian, tubal or peritoneal cancers
Enrollment: 12 (Actual)
Dates: Start 2021-05-05 (Actual); Primary Completion 2025-04-17 (Actual); Study Completion 2025-04-17 (Actual)

PRIMARY OUTCOMES:
Identification of metrics (clinical, biological, pharmacokinetic) that are considered as toxicity induction causes (hematological toxicity or nephrotoxicity) | Month 10; after all the blood sample collection is achieved for all included patients.
  Blood will be sampled at Cycle 1 Day 1, Cycle 1 Day 15, Cycle 2 Day 1 and Cycle 3 Day 1 and based on the obtained results, it will be seek if a link can be established between the clinical, biological and pharmacokinetic metrics and the observed toxicity.

SECONDARY OUTCOMES:
Determination of the average pharmacokinetic metrics observed in our study panel patients. | Month 10; after all the blood sample collection is achieved for all included patients..
  Blood will be sampled at Cycle 1 Day 1, Cycle 1 Day 15, Cycle 2 Day 1 and Cycle 3 Day 1 and based on the obtained results, the average metrics of pharmacokinetic parameters will be determined.
Relationship between the pharmacokinetic metrics and the PFS at 24 months. | Month 34; after last patient inclusion (Month 10) + 24 months.
  Blood will be sampled at Cycle 1 Day 1, Cycle 1 Day 15, Cycle 2 Day 1 and Cycle 3 Day 1 and based on the obtained results, it will be determined if a link can be established between the pharmacokinetic metrics and the PFS at 24 months
Relationship between the quality of life and the observed toxicity assessed by the "EORTC OVARIAN" questionnaire | Month 10, after last patient enrolment.
  Analysis of quality of life by "QLQ OV28" questionnaire score collected at Cycle 1 Day 1, Cycle 1 Day 15, Cycle 2 Day 1 and Cycle 3 Day 1 and observed toxicity.
Relationship between the quality of life and the observed toxicity assessed by the "Charlson Score" questionnaire | Month 10, after last patient enrolment.
  Analysis of quality of life by "Charlson Score" questionnaire score collected at Cycle 1 Day 1, Cycle 1 Day 15, Cycle 2 Day 1 and Cycle 3 Day 1 and observed toxicity.
Relationship between the quality of life and the observed toxicity assessed by the "Assessment of polymedication" questionnaire | Month 10, after last patient enrolment.
  Analysis of quality of life by "Assessment of polymedication" questionnaire score collected at Cycle 1 Day 1, Cycle 1 Day 15, Cycle 2 Day 1 and Cycle 3 Day 1 and observed toxicity.
Relationship between the quality of life and the observed toxicity assessed by the "Recording of food intake and monitoring of eating habits" questionnaire | Month 10, after last patient enrolment.
  Analysis of quality of life by "Recording of food intake and monitoring of eating habits" questionnaire score collected at Cycle 1 Day 1, Cycle 1 Day 15, Cycle 2 Day 1 and Cycle 3 Day 1 and observed toxicity.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Lyon sud, Institut de Cancérologie des Hospices Civils de Lyon, Pierre-Bénite, France

IPD SHARING:
Plan to Share IPD: No